CLINICAL TRIAL: NCT03062969
Title: The Transition From Blastomere to Trophectoderm Biopsy: Comparing Two PGS Strategies
Status: Completed | Type: Observational
Sponsor: Fundacion Dexeus (Other)
Responsible Party: Principal Investigator, Lluc Coll Lujan, Principal investigator, Fundacion Dexeus
Other Study IDs: FDS-PGS-01
Record Dates: First submitted 2017-02-16; First posted 2017-02-24 (Actual); Last update posted 2017-02-24 (Actual); Status verified 2017-02

CONDITIONS: Infertility; Preimplantation Genetic Screening
MeSH Terms: conditions — Infertility

STUDY DESIGN:
Observational Model: Case-Crossover | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Cleavage stage biopsy group: Patients undergoing a PGS cycle with single blastomere biopsy on day 3 and analysis using comparative genomic hybridation bacterial artificial chromosome (BAC) arrays (aCGH) If euploid blastocysts were available, patients underwent fresh blastocyst transfer on day 5.
  Interventions: Procedure: Cleavage stage biopsy group
- Trophectoderm biopsy group: Patients undergoing a PGS cycle with blastocyst biopsy on day 5-7 and analysis using comparative genomic hybridation bacterial artificial chromosome (BAC) arrays (aCGH). If euploid blastocysts were available, patients underwent frozen-thawed blastocyst transfer.
  Interventions: Procedure: Trophectoderm biopsy group

INTERVENTIONS:
Procedure: Cleavage stage biopsy group — * intracytoplasmatic sperm injection (ICSI)- (Invitro Fertilization)IVF
  * Time lapse embryo culture
  * Cleavage stage biopsy
  * aCGH analysis
  * Fresh euploid embryo transfer
  Groups: Cleavage stage biopsy group
Procedure: Trophectoderm biopsy group — * ICSI-IVF
  * Time lapse embryo culture
  * Day 3 zona pellucida opening
  * Trophectoderm biopsy
  * aCGH analysis
  * Frozen-thawed euploid embryo transfer
  Groups: Trophectoderm biopsy group

SUMMARY:
Shortly after the implementation of Comprehensive Chromosome Screening (CCS) techniques for Preimplantation Genetic Screening (PGS) came the transition in biopsy timing. Trophectoderm biopsy is meant to overcome the limitations of cleavage stage biopsy and single cell analysis.

DETAILED DESCRIPTION:
The investigators have recently introduced this new approach and a frozen-thawed policy of euploid blastocysts is routinely performed.

This is a single centre retrospective study in patients undergoing a PGS cycle. The aim of the study is to assess the results obtained in a PGS programme after the implementation of a new biopsy timing and transfer policy. Results obtained in PGS cycles with blastocyst biopsy and frozen-thawed embryo transfer were analysed in comparison to cycles with cleavage stage biopsy and fresh blastocyst transfer.

ELIGIBILITY:
Inclusion Criteria:

* Own gametes
* PGS for: advanced maternal age, repeated implantation failure, recurrent miscarriages, severe male factor, and previous affected pregnancies

Exclusion Criteria:

* PGS cycles with gamete donation
* Altered karyotypes
* Combined Preimplantation genetic diagnosis (PGD)+PGS cycles

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Study Population: Patients undergoing a PGS cycle with own gametes for any of the following indications: advanced maternal age, repeated implantation failure, recurrent miscarriages, severe male factor, and previous affected pregnancies.
Sampling Method: Non-Probability Sample
Enrollment: 383 (Actual)
Dates: Start 2014-01-01 (Actual); Primary Completion 2016-02-28 (Actual); Study Completion 2017-01 (Actual)

PRIMARY OUTCOMES:
Ongoing clinical pregnancy rate | 20 weeks after embryo transfer
  Clinical pregnancy confirmed by ultrasound

SECONDARY OUTCOMES:
Implantation Rate | 6 weeks after embryo transfer
  Embryos implanted confirmed by ultrasound
Number of available euploid blastocysts per cycle | Up to 15 days after embryo biopsy
  Transferable or vitrified euploid blastocysts
Miscarriage Rate | Until 20 weeks after embryo transfer

IPD SHARING:
Plan to Share IPD: No